CLINICAL TRIAL: NCT04088734
Title: A Phase I/II Open Label, Single-dose, Gene Transfer Study of scAAV9.U1a.hSGSH (ABO-102) in Patients With Middle and Advanced Phases of MPS IIIA Disease
Brief Title: Gene Transfer Study of ABO-102 in Patients With Middle and Advanced Phases of MPS IIIA Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to lack of efficacy seen in patients with advanced MPS IIIA disease. The patients will be followed up annually for safety until five years post dosing
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Collaborators: Abeona Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-003; UX111-CL201 (Other: Ultragenyx Pharmaceutical Inc); 2018-000504-42 (EudraCT Number)
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Results first posted 2023-07-25 (Actual); Last update posted 2023-07-25 (Actual); Status verified 2023-07

CONDITIONS: MPS IIIA; Sanfilippo Syndrome; Sanfilippo A; Mucopolysaccharidosis III
Keywords: MPS IIIA; Sanfilippo; Gene therapy
MeSH Terms: conditions — Mucopolysaccharidosis III

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABO-102 (Experimental): Dose of 3x10^13 vg/kg
  Interventions: Drug: ABO-102

INTERVENTIONS:
Drug: ABO-102 — Single dose of ABO-102 (scAAV9.U1a.hSGSH) administered by intravenous injection through a peripheral limb vein at a dose of 3 X 10^13 vg/kg
  Other Names: scAAV9.U1a.hSGSH; UX111

SUMMARY:
Open-label, clinical trial of scAAV9.U1a.hSGSH injected intravenously through a peripheral limb vein

DETAILED DESCRIPTION:
This is an open-label, single dose clinical trial. All participants will receive 3 X 10^13 vg/kg of ABO-102 delivered one time through a venous catheter inserted into a peripheral limb vein. The target population includes MPS IIIA participants with a DQ lower than 60 in middle and advanced phases of the disease. Similar numbers of MPS IIIA participants with age equivalent above and below 18 months of age will be enrolled to ensure a representation of middle and advanced phases of the disease.

This study was previously posted by Abeona Therapeutics, Inc and was transferred to Ultragenyx in August 2022.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MPS IIIA confirmed by the following methods:

  1. No detectable or significantly reduced SGSH enzyme activity by leukocyte assay and
  2. Genomic DNA analysis demonstrating homozygous or compound heterozygous mutations in the SGSH gene
* Cognitive Development Quotient (DQ) lower than 60 (calculated by Bayley Scales of Infant and Toddler Development - Third Edition)
* Must be ambulatory, though may receive assistance with ambulation
* Age range of 2 years up to 18 years (excluded)

Exclusion Criteria:

* Inability to participate in the clinical evaluation as determined by Principal Investigator
* Identification of two nonsense or null variants on genetic testing of the SGSH gene
* At least one S298P mutation in the SGSH gene
* Has evidence of an attenuated phenotype of MPS IIIA
* Presence of a concomitant medical condition that precludes lumbar puncture or use of anesthetics
* Active viral infection based on clinical observations
* Concomitant illness or requirement for chronic drug treatment that in the opinion of the PI creates unnecessary risks for gene transfer, or precludes the child from participating in the protocol assessments and follow up
* Participants with total anti-AAV9 antibody titers greater than or equal to 1:100 as determined by ELISA binding immunoassay
* Participants with a positive response for the ELISPOT for T-cell responses to AAV9
* Serology consistent with exposure to HIV, or serology consistent with active hepatitis B or C infection
* Bleeding disorder or any other medical condition or circumstance in which a lumbar puncture (for collection of CSF) is contraindicated according to local institutional policy
* Visual or hearing impairment sufficient to preclude cooperation with neurodevelopmental testing
* Any item (braces, etc.) which would exclude the participant from being able to undergo MRI according to local institutional policy
* Any other situation that precludes the participant from undergoing procedures required in this study
* Participants with cardiomyopathy or significant congenital heart abnormalities
* The presence of significant non-MPS IlIA related CNS impairment or behavioral disturbances that would confound the scientific rigor or interpretation of results of the study
* Abnormal laboratory values Grade 2 or higher as defined in CTCAE v4.03 for GGT, total bilirubin (except in subjects diagnosed with Gilbert's syndrome), creatinine, hemoglobin, WBC count, platelet count, PT and aPTT
* Female participant who is pregnant or demonstrates a positive urine or beta-hCG result at screening assessment (if applicable)
* Any vaccination with viral attenuated vaccines less than 30 days prior to the scheduled date of treatment (and use of prednisolone)
* Previous treatment by Haematopoietic Stem Cell transplantation
* Previous participation in a gene/cell therapy or ERT clinical trial
* Participants who are anticipated to undergo a procedure involving anesthesia within 6 months post- drug administration
* Dysphagia present at Grade 3 or higher, as defined in CTCAE v4.03

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2022-03-10 (Actual); Study Completion 2022-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (3):
- Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States
- Adelaide Women's and Children's Hospital, North Adelaide, South Australia, Australia
- Hospital Clínico Universitario de Santiago, Santiago de Compostela, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fu H, Cataldi MP, Ware TA, Zaraspe K, Meadows AS, Murrey DA, McCarty DM. Functional correction of neurological and somatic disorders at later stages of disease in MPS IIIA mice by systemic scAAV9-hSGSH gene delivery. Mol Ther Methods Clin Dev. 2016 Jun 8;3:16036. doi: 10.1038/mtm.2016.36. eCollection 2016. PMID 27331076
- [Background] Fu H, Meadows AS, Pineda RJ, Kunkler KL, Truxal KV, McBride KL, Flanigan KM, McCarty DM. Differential Prevalence of Antibodies Against Adeno-Associated Virus in Healthy Children and Patients with Mucopolysaccharidosis III: Perspective for AAV-Mediated Gene Therapy. Hum Gene Ther Clin Dev. 2017 Dec;28(4):187-196. doi: 10.1089/humc.2017.109. Epub 2017 Oct 24. PMID 29064732

RESULTS

PARTICIPANT FLOW:
Groups:
- scAAV9.U1a.hSGSH, 3x1013 vg/kg: An intravenous injection of ABO-102 (scAAV9.U1a.hSGSH) via peripheral limb vein at a dose of 3.0 x 1013 vg/kg
Period: Overall Study
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Started | 5
Completed | 0
Not Completed | 5
Not completed — Other, Not Specified | 5

BASELINE CHARACTERISTICS:
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: months] | 69.02 (34.692)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 5

OUTCOME MEASURES:

1. Primary Outcome: Incidence, Type and Severity of Related Treatment-Emergent Adverse Events (TEAEs) by Time Frame
Description: An adverse event (AE) is any untoward medical occurrence or unintended change from the time informed consent form (ICF) is signed, including inter-current illness that occurs during the course of a clinical trial after treatment has started, whether considered related to treatment or not. TEAEs are those that occurred after the start of study drug. Related adverse events were categorized as possible, probable, or definitely.
Time Frame: From the first dose of study drug to <30 days postdose, Day 30, 60, 90, 180 and Month 12
Measure: Number; unit: participants
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 5
participants
  < 30 days : Possible; Mild | 1
  < 30 days : Possible; Moderate | 0
  < 30 days : Possible; Severe | 0
  < 30 days : Probable; Mild | 2
  < 30 days : Probable; Moderate | 0
  < 30 days : Probable; Severe | 1
  < 30 days : Definitely; Mild | 1
  < 30 days : Definitely; Moderate | 0
  < 30 days : Definitely; Severe | 0
  30 - < 60 days : Possible; Mild | 0
  30 - < 60 days : Possible; Moderate | 0
  30 - < 60 days : Possible; Severe | 0
  30 - < 60 days : Probable; Mild | 2
  30 - < 60 days : Probable; Moderate | 0
  30 - < 60 days : Probable; Severe | 1
  30 - < 60 days : Definitely; Mild | 1
  30 - < 60 days : Definitely; Moderate | 0
  30 - < 60 days : Definitely; Severe | 0
  60 - < 90 days : Possible; Mild | 0
  60 - < 90 days : Possible; Moderate | 0
  60 - < 90 days : Possible; Severe | 0
  60 - < 90 days : Probable; Mild | 1
  60 - < 90 days : Probable; Moderate | 0
  60 - < 90 days : Probable; Severe | 0
  60 - < 90 days : Definitely; Mild | 0
  60 - < 90 days : Definitely; Moderate | 0
  60 - < 90 days : Definitely; Severe | 0
  90 - < 180 days : Possible; Mild | 0
  90 - < 180 days : Possible; Moderate | 0
  90 - < 180 days : Possible; Severe | 0
  90 - < 180 days : Probable; Mild | 0
  90 - < 180 days : Probable; Moderate | 1
  90 - < 180 days : Probable; Severe | 0
  90 - < 180 days : Definitely; Mild | 0
  90 - < 180 days : Definitely; Moderate | 0
  90 - < 180 days : Definitely; Severe | 0
  180 - < 12 months : Possible; Mild | 0
  180 - < 12 months : Possible; Moderate | 0
  180 - < 12 months : Possible; Severe | 1
  180 - < 12 months : Probable; Mild | 0
  180 - < 12 months : Probable; Moderate | 0
  180 - < 12 months : Probable; Severe | 0
  180 - < 12 months : Definitely; Mild | 0
  180 - < 12 months : Definitely; Moderate | 0
  180 - < 12 months : Definitely; Severe | 0

2. Primary Outcome: Incidence, Type and Severity of Serious Adverse Events (SAEs) by Time Frame
Description: An SAE is defined as any untoward medical occurrence that, at any dose:
  1. Results in death
  2. Is life threatening
  3. Requires inpatient hospitalization or prolongation of existing hospitalization
  4. Results in persistent disability/incapacity
  5. Is a congenital anomaly/birth defect
  6. Other situations such as important medical events that may not be immediately life threatening or result in death or hospitalization but may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition.
  Relationship to study drug was defined as unrelated, unlikely, possible, probable, or definitely.
Time Frame: From signing of informed consent through Day 60, 90, 180 and up to Day 454 (> 12 months)
Measure: Count of Participants; unit: Participants
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 5
Participants
  60 - < 90 days : Unrelated; Mild | 0
  60 - < 90 days : Unrelated; Moderate | 0
  60 - < 90 days : Unrelated; Severe | 0
  60 - < 90 days : Unlikely; Mild | 0
  60 - < 90 days : Unlikely; Moderate | 0
  60 - < 90 days : Unlikely; Severe | 1
  60 - < 90 days : Possible; Mild | 0
  60 - < 90 days : Possible; Moderate | 0
  60 - < 90 days : Possible; Severe | 0
  60 - < 90 days : Probable; Mild | 0
  60 - < 90 days : Probable; Moderate | 0
  60 - < 90 days : Probable; Severe | 0
  60 - < 90 days : Definite; Mild | 0
  60 - < 90 days : Definite; Moderate | 0
  60 - < 90 days : Definite; Severe | 0
  90 - < 180 days : Unrelated; Mild | 0
  90 - < 180 days : Unrelated; Moderate | 0
  90 - < 180 days : Unrelated; Severe | 1
  90 - < 180 days : Unlikely; Mild | 0
  90 - < 180 days : Unlikely; Moderate | 0
  90 - < 180 days : Unlikely; Severe | 1
  90 - < 180 days : Possible; Mild | 0
  90 - < 180 days : Possible; Moderate | 0
  90 - < 180 days : Possible; Severe | 0
  90 - < 180 days : Probable; Mild | 0
  90 - < 180 days : Probable; Moderate | 0
  90 - < 180 days : Probable; Severe | 0
  90 - < 180 days : Definite; Mild | 0
  90 - < 180 days : Definite; Moderate | 0
  90 - < 180 days : Definite; Severe | 0
  180 days - < 12 months : Unrelated; Mild | 0
  180 days - < 12 months : Unrelated; Moderate | 0
  180 days - < 12 months : Unrelated; Severe | 0
  180 days - < 12 months : Unlikely; Mild | 0
  180 days - < 12 months : Unlikely; Moderate | 0
  180 days - < 12 months : Unlikely; Severe | 0
  180 days - < 12 months : Possible; Mild | 0
  180 days - < 12 months : Possible; Moderate | 0
  180 days - < 12 months : Possible; Severe | 1
  180 days - < 12 months : Probable; Mild | 0
  180 days - < 12 months : Probable; Moderate | 0
  180 days - < 12 months : Probable; Severe | 0
  180 days - < 12 months : Definite; Mild | 0
  180 days - < 12 months : Definite; Moderate | 0
  180 days - < 12 months : Definite; Severe | 0
  >= 12 months : Unrelated; Mild | 0
  >= 12 months : Unrelated; Moderate | 0
  >= 12 months : Unrelated; Severe | 1
  >= 12 months : Unlikely; Mild | 0
  >= 12 months : Unlikely; Moderate | 0
  >= 12 months : Unlikely; Severe | 0
  >= 12 months : Possible; Mild | 0
  >= 12 months : Possible; Moderate | 0
  >= 12 months : Possible; Severe | 0
  >= 12 months : Probable; Mild | 0
  >= 12 months : Probable; Moderate | 0
  >= 12 months : Probable; Severe | 0
  >= 12 months : Definite; Mild | 0
  >= 12 months : Definite; Moderate | 0
  >= 12 months : Definite; Severe | 0

3. Primary Outcome: Change From Baseline (BL) in Multiples of Normal of Liver and Spleen Volumes After Treatment
Description: As Measured by Magnetic Resonance Imaging (MRI). Baseline value of multiple of normal is calculated using the baseline values of the Liver volume/Spleen Volume/Height and Weight.
  * Body Surface Area (BSA) (m2)=( Height(cm) * Weight (kg)/3600)1/2.
  * Normal Liver Volume=(689.9 * BSA (m)) - 24.7.
  * Normal Spleen Volume (mL)=(4.6 * Weight (kg)) + 0.7.
  * Liver Volume (multiples of normal)=Subject Liver Volume (mL)/Normal Liver Volume (mL).
  * Spleen Volume (multiples of normal)=Subject Spleen Volume (mL)/Normal Spleen Volume (mL).
Time Frame: Baseline, Day 30, 180, Month 12
Population: Participants with an assessment at baseline and given time point
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 5
ratio
  Liver volume: change from BL to Day 30: number analyzed (Participants) | 3
  Liver volume: change from BL to Day 30 | -0.4200 (0.08876)
  Liver volume: change from BL to Day 180: number analyzed (Participants) | 3
  Liver volume: change from BL to Day 180 | -0.4543 (0.31560)
  Liver volume: change from BL to Month 12: number analyzed (Participants) | 2
  Liver volume: change from BL to Month 12 | -0.1765 (0.17466)
  Spleen volume: change from BL to Day 30: number analyzed (Participants) | 4
  Spleen volume: change from BL to Day 30 | -0.0603 (0.19257)
  Spleen volume: change from BL to Day 180: number analyzed (Participants) | 3
  Spleen volume: change from BL to Day 180 | -0.2253 (0.53267)
  Spleen volume: change from BL to Month 12: number analyzed (Participants) | 2
  Spleen volume: change from BL to Month 12 | -0.1330 (0.18102)

4. Primary Outcome: Change From BL in Cerebrospinal Fluid (CSF) Heparan Sulfate Levels After Treatment
Description: Change from baseline in CSF heparan sulfate levels after treatment
Time Frame: Baseline, Day 30, Day 180, Month 12
Population: Participants with an assessment at given time point
Measure: Mean (Standard Deviation); unit: nmol/mL
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 5
nmol/mL
  Change from BL to Day 30 | -0.120 (0.0837)
  Change from BL to Day 180: number analyzed (Participants) | 3
  Change from BL to Day 180 | -0.183 (0.0289)
  Change from BL to Month 12: number analyzed (Participants) | 1
  Change from BL to Month 12 | -0.100 (NA) — 1 participant analyzed

5. Secondary Outcome: Change From Baseline in Plasma Heparan Sulfate After Treatment
Time Frame: Baseline, Day 30, Day 180, Month 12
Population: Participants with an assessment at given time point
Measure: Mean (Standard Deviation); unit: pmol/mL
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 5
pmol/mL
  Change from Baseline to Day 30 | -31.0 (9.62)
  Change from Baseline to Day 180: number analyzed (Participants) | 4
  Change from Baseline to Day 180 | -25.0 (7.07)
  Change from Baseline to Month 12: number analyzed (Participants) | 2
  Change from Baseline to Month 12 | -17.5 (17.68)

6. Secondary Outcome: Change From Baseline in Urine Glycosaminoglycans After Treatment
Time Frame: Baseline, Day 30, Day 180, Month 12
Population: Participants with an assessment at given time point
Measure: Mean (Standard Deviation); unit: mg/mmol creatinine
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 5
mg/mmol creatinine
  Change from Baseline to Day 30: number analyzed (Participants) | 4
  Change from Baseline to Day 30 | -14.5 (9.33)
  Change from Baseline to Day 180: number analyzed (Participants) | 3
  Change from Baseline to Day 180 | -13.7 (9.81)
  Change from Baseline to Month 12: number analyzed (Participants) | 1
  Change from Baseline to Month 12 | -4.0 (NA) — 1 participant analyzed

7. Secondary Outcome: Change From Baseline in Urine Heparan Sulfate After Treatment
Time Frame: Baseline, Day 30, Day 180, Month 12
Population: Participants with an assessment at given time point
Measure: Mean (Standard Deviation); unit: μmol/mmol creatinine
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 5
μmol/mmol creatinine
  Change from Baseline to Day 30: number analyzed (Participants) | 4
  Change from Baseline to Day 30 | -0.95 (0.676)
  Change from Baseline to Day 180: number analyzed (Participants) | 3
  Change from Baseline to Day 180 | -0.63 (0.651)
  Change from Baseline to Month 12: number analyzed (Participants) | 1
  Change from Baseline to Month 12 | 0.60 (NA) — 1 participant analyzed

8. Secondary Outcome: Change From Baseline in CSF N-Sulfoglucosamine Sulfohydrolase (SGSH) Enzyme Activity Levels After Treatment
Time Frame: Baseline, Day 30, Day 180, and Month 12
Population: Participants with an assessment at given time point
Measure: Mean (Standard Deviation); unit: nmol/17 h/mL
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 5
nmol/17 h/mL
  Change from Baseline to Day 30 | 2.662 (5.9524)
  Change from Baseline to Day 180: number analyzed (Participants) | 3
  Change from Baseline to Day 180 | -3.297 (5.7100)
  Change from Baseline to Month 12: number analyzed (Participants) | 1
  Change from Baseline to Month 12 | 0.000 (NA) — 1 participant analyzed

9. Secondary Outcome: Change From Baseline in Heparan N-Sulfatase (Type A) After Treatment
Time Frame: Baseline, Day 30, Day 180, Month 12
Population: Participants with an assessment at given time point
Measure: Mean (Standard Deviation); unit: nmol/17 h/mL
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 5
nmol/17 h/mL
  Change from Baseline to Day 30 | 0.578 (1.1299)
  Change from Baseline to Day 180: number analyzed (Participants) | 3
  Change from Baseline to Day 180 | 0.000 (0.0000)
  Change from Baseline to Month 12: number analyzed (Participants) | 2
  Change from Baseline to Month 12 | 0.025 (0.0354)

10. Secondary Outcome: Change From Baseline in Plasma SGSH After Treatment
Time Frame: Baseline, Day 30, Day 180, Month 12
Population: Participants with an assessment at given time point
Measure: Mean (Standard Deviation); unit: nmol/17 h/mL
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 5
nmol/17 h/mL
  Change from Baseline to Day 30 | 6.50 (8.682)
  Change from Baseline to Day 180: number analyzed (Participants) | 4
  Change from Baseline to Day 180 | 0.88 (1.825)
  Change from Baseline to Month 12: number analyzed (Participants) | 2
  Change from Baseline to Month 12 | 0.05 (0.495)

11. Secondary Outcome: Change From Baseline in Brain Volumes After Treatment
Description: As measured by MRI
Time Frame: Baseline, 12 months
Population: Participants with an assessment
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 2
mL
  Change in amygdala volume | -0.635 (0.2333)
  Change in corpus callosum volume | 0.285 (0.5445)
  Change in CSF volume | 1.290 (0.5091)
  Change in total cerebellar gray matter volume | -7.210 (7.2125)
  Change in total cerebellar white matter volume | 0.985 (4.0234)
  Change in total brain volume | -157.705 (44.6114)
  Change in total cerebral volume | -152.365 (59.1353)
  Change in total cerebral gray matter volume | -145.975 (81.0981)
  Change in total cortical volume | -144.170 (84.9235)
  Change in total cerebellar volume | -6.225 (11.2218)
  Change in total cerebral white matter volume | -6.385 (21.9698)
  Change in total gray matter volume | -153.190 (73.8927)
  Change in total intercranial volume | -122.245 (40.0576)
  Change in total white matter volume | -5.400 (25.9932)
  Change in ventricular volumes | 34.165 (5.0417)

12. Secondary Outcome: Change From Baseline in Brain Volumes After Treatment: Average Total Cortical Thickness
Description: As measured by MRI
Time Frame: Baseline, 12 months
Population: Participants with an assessment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 2
mm | -0.455 (0.2475)

13. Secondary Outcome: Change From Baseline in Sleep Pattern as Measured by the Modified Children's Sleep Habits Questionnaire (CSHQ) Subscore Total After Treatment
Description: CSHQ is a caregiver-completed, 35-item questionnaire that assesses the frequency of behaviors associated with common pediatric sleep difficulties. Eight domains of sleep, including Bedtime Resistance, Sleep Onset Delay, Sleep Duration, Sleep Anxiety, Night Awakenings, Parasomnias, Sleep Disordered Breathing, and Daytime Sleepiness are assessed, producing eight individual subdomain scores and an overall CSHQ subscore total. CSHQ total score is calculated by adding all the 8 subscores, and ranges from 36 to 108. A higher score is indicative of more disturbed sleep.
Time Frame: Baseline, Day 180, Month 12
Population: participants with an assessment at given time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 5
score on a scale
  Change from Baseline to Day 180 | 2.8 (4.76)
  Change from Baseline to Month 12: number analyzed (Participants) | 2
  Change from Baseline to Month 12 | 1.5 (3.54)

14. Secondary Outcome: Change From Baseline in Pediatric Quality of Life Inventory (PedsQL™) Core Generic Scales Total Score
Description: PedsQL is a brief measure of health-related quality of life in children. The Peds QL Generic Core Scales was used in the study, consisting of 23 items applicable for healthy school and community populations, as well as pediatric populations with acute and chronic conditions. The four scales include Physical Functioning, Emotional Functioning, Social Functioning, and School Functioning. Item scores are added together and averaged to produce a Core total score, where higher scores on a scale of 0-100 indicate better Health-related Quality of Life (HRQOL).
Time Frame: Baseline, Day 180, Month 12
Population: Participants with an assessment at given time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 5
score on a scale
  Change from Baseline to Day 180 | -11.60 (23.218)
  Change from Baseline to Month 12: number analyzed (Participants) | 2
  Change from Baseline to Month 12 | -23.80 (6.647)

15. Secondary Outcome: Change From Baseline in Parent Quality of Life, Using the Parenting Stress Index, 4th Edition (PSI-4) Total Stress Raw Score
Description: The Parenting Stress Index, 4th Edition evaluates the magnitude and type of stress in a parent/child relationship. The short form version was used in the study, consisting of 36 items divided into three domains: Parental Distress (PD), Parent-Child Dysfunctional Interaction (P-CDI), and Difficult Child (DC), which combine together to form a Total Stress raw score. Total Stress raw scores can range from 36 - 180, with higher raw scores indicating higher levels of stress.
Time Frame: Baseline, Day 180, Month 12
Population: Participants with an assessment at given time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 5
score on a scale
  Change from Baseline to Day 180: number analyzed (Participants) | 3
  Change from Baseline to Day 180 | -14.0 (24.33)
  Change from Baseline to Month 12: number analyzed (Participants) | 2
  Change from Baseline to Month 12 | -9.0 (4.24)

16. Secondary Outcome: Change From Baseline in Gastrointestinal Symptoms Using the PedsQL™ Gastrointestinal (GI) Symptoms Scales Score
Description: The PedsQL Gastrointestinal Symptoms Scale is a specific module of the PedsQL that measures gastrointestinal symptoms in patients with acute and chronic health conditions as well as healthy school and community populations. The Parent Report version was used on the study, consisting of 58 items across 10 dimensions, assessing parents' perceptions of their child's GI-specific symptoms. Item scores are added together and averaged to produce a GI symptoms scales score, where higher scores on a scale of 0-100 indicate better GI specific QOL.
Time Frame: Baseline, Day 180, Month 12
Population: Participants with an assessment at given time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 5
score on a scale
  Change from Baseline to Day 180: number analyzed (Participants) | 4
  Change from Baseline to Day 180 | -5.88 (9.261)
  Change from Baseline to Month 12: number analyzed (Participants) | 2
  Change from Baseline to Month 12 | -4.15 (6.010)

17. Secondary Outcome: Change From Baseline in Parent Global Impression (PGI) Total Score
Description: The Parent Global Impression scale evaluates all aspects of a patients' health and assesses if there has been an improvement or decline in clinical status, as reported by the parent/caregiver. This study used a modified version with symptoms relevant to the patient population in the trial. Nine symptoms were scored at each visit, using a 7-point rating scale where 3 = much better, 2 = better, 1 = slightly better, 0 = same, -1 = slightly worse, -2 = worse, and -3 = much worse. The nine symptom scores are added together to produce a PGI total score, ranging from -27 to 27.
Time Frame: Baseline, Day 180, Month 12
Population: Participants with an assessment at given time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 5
score on a scale
  Change at Day 180: number analyzed (Participants) | 4
  Change at Day 180 | -3.0 (6.48)
  Change at Month 12: number analyzed (Participants) | 3
  Change at Month 12 | -3.0 (6.56)

18. Secondary Outcome: Clinical Global Impression Improvement Scale at Day 180 and Month 12
Description: The Clinical Global Impression of Improvement scale is a brief, stand-alone assessment of the clinician's view of the patient's global functioning prior to and after initiating a study medication, specifically looking at whether the patient has demonstrated improvement or not. Assessment of improvement was scored at each visit, using a 7-point rating scale where 0 = not assessed, 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse.
Time Frame: Day 180, Month 12
Population: Participants with an assessment at given time point
Measure: Count of Participants; unit: Participants
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 5
Participants
  Global Improvement, Day 180: number analyzed (Participants) | 4
  Global Improvement, Day 180: 0 = not assessed | 0
  Global Improvement, Day 180: 1 = very much improved | 0
  Global Improvement, Day 180: 2 = much improved | 0
  Global Improvement, Day 180: 3 = minimally improved | 0
  Global Improvement, Day 180: 4 = no change | 1
  Global Improvement, Day 180: 5 = minimally worse | 1
  Global Improvement, Day 180: 6 = much worse | 2
  Global Improvement, Day 180: 7 = very much worse | 0
  Global Improvement, Month 12: number analyzed (Participants) | 3
  Global Improvement, Month 12: 0 = not assessed | 0
  Global Improvement, Month 12: 1 = very much improved | 0
  Global Improvement, Month 12: 2 = much improved | 0
  Global Improvement, Month 12: 3 = minimally improved | 1
  Global Improvement, Month 12: 4 = no change | 0
  Global Improvement, Month 12: 5 = minimally worse | 0
  Global Improvement, Month 12: 6 = much worse | 2
  Global Improvement, Month 12: 7 = very much worse | 0

19. Secondary Outcome: Change From Baseline in Parent Symptoms Score Questionnaire
Description: The Parent Symptoms Score Questionnaire contains 29 symptoms with an indicator of whether the symptom was present or absent.
Time Frame: Baseline, Day 180, Month 12
Population: Due to the inconsistent use of forms across visits and sites for this study, the data collected for this endpoint was incomplete, unreliable, and could not be evaluated.
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 0

20. Secondary Outcome: Percent Change From Baseline in Body Mass Index After Treatment
Time Frame: Baseline, Day 30, Day 180, Month 12
Population: Participants with an assessment at given time point
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 5
percent change
  Change from Baseline to Day 30: number analyzed (Participants) | 4
  Change from Baseline to Day 30 | -0.581 (4.4477)
  Change from Baseline to Day 180: number analyzed (Participants) | 3
  Change from Baseline to Day 180 | 3.875 (9.0517)
  Change from Baseline to Month 12: number analyzed (Participants) | 2
  Change from Baseline to Month 12 | 9.873 (6.1672)

21. Secondary Outcome: Number of Participants With Abnormalities in Standard Awake 45-Minutes-Electroencephalogram (EEG) Monitoring at Baseline and Day 180
Description: NCS=not clinically significant CS=clinically significant
Time Frame: Baseline, Day 180
Population: Participants with an assessment
Measure: Count of Participants; unit: Participants
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 3
Participants
  Overall EEG : Baseline: Abnormal, CS | 0
  Overall EEG : Baseline: Abnormal, NCS | 3
  Overall EEG : Baseline: Normal | 0
  Overall EEG : Day 180: Abnormal, CS | 1
  Overall EEG : Day 180: Abnormal, NCS | 1
  Overall EEG : Day 180: Normal | 1

22. Secondary Outcome: Change From Baseline in Vector Shedding Analysis in Plasma, Saliva, Stool and Urine
Description: Detection of the adeno-associated Virus 9 (AAV9) viral deoxyribonucleic acid (DNA) in plasma, saliva, urine and feces was analyzed. Per protocol, data were not collected for urine at Month 12.
Time Frame: Baseline, Day 30, Day 180, Month 12
Population: Participants with an assessment at given time point
Measure: Mean (Standard Deviation); unit: Copies per 1 mL of Specimen (copies/mL)
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
Number analyzed (Participants) | 5
Copies per 1 mL of Specimen (copies/mL)
  Plasma Change from Baseline to Day 30 | 45115.0 (45413.33)
  Plasma Change from Baseline to Day 180: number analyzed (Participants) | 4
  Plasma Change from Baseline to Day 180 | -2686.3 (5372.50)
  Plasma Change from Baseline to Month 12: number analyzed (Participants) | 2
  Plasma Change from Baseline to Month 12 | 2250.0 (3181.98)
  Saliva Change from Baseline to Day 30: number analyzed (Participants) | 2
  Saliva Change from Baseline to Day 30 | 17472.5 (18345.89)
  Saliva Change from Baseline to Day 180: number analyzed (Participants) | 3
  Saliva Change from Baseline to Day 180 | -1900.3 (2330.09)
  Saliva Change from Baseline to Month 12: number analyzed (Participants) | 1
  Saliva Change from Baseline to Month 12 | 0.0 (NA) — Not applicable; 1 participant analyzed
  Stool Change from Baseline to Day 30: number analyzed (Participants) | 4
  Stool Change from Baseline to Day 30 | -277522.5 (760910.43)
  Stool Change from Baseline to Day 180: number analyzed (Participants) | 2
  Stool Change from Baseline to Day 180 | -800833.0 (1132548.89)
  Stool Change from Baseline to Month 12: number analyzed (Participants) | 1
  Stool Change from Baseline to Month 12 | 0.0 (NA) — Not applicable; 1 participant analyzed
  Urine Change from Baseline to Day 30: number analyzed (Participants) | 4
  Urine Change from Baseline to Day 30 | 2250.0 (2598.08)
  Urine Change from Baseline to Day 180: number analyzed (Participants) | 3
  Urine Change from Baseline to Day 180 | 1500.0 (2598.08)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: From enrollment to the end of study; mean of 18 months. Adverse Events: from first dose of study drug up to Day 454.
Arm/Group | scAAV9.U1a.hSGSH, 3x1013 vg/kg
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | scAAV9.U1a.hSGSH, 3x1013 vg/kg (N=5)
Dysphagia (Gastrointestinal disorders) | 1
Gait disturbance (General disorders) | 1
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 1
Cognitive disorder (Nervous system disorders) | 2
Mental status changes (Psychiatric disorders) | 1
Gastrostomy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | scAAV9.U1a.hSGSH, 3x1013 vg/kg (N=5)
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Mixed deafness (Ear and labyrinth disorders) | 1
Cushingoid (Endocrine disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 4
Gait disturbance (General disorders) | 1
Cellulitis (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 3
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 5
Blood creatine phosphokinase increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 3
Haematocrit increased (Investigations) | 1
Haemoglobin increased (Investigations) | 1
Platelet count decreased (Investigations) | 1
Red blood cell count increased (Investigations) | 1
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Dyskinesia (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Fine motor skill dysfunction (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Abnormal behaviour (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 1
Initial insomnia (Psychiatric disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/34/NCT04088734/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-15): https://cdn.clinicaltrials.gov/large-docs/34/NCT04088734/SAP_001.pdf